CLINICAL TRIAL: NCT03125941
Title: Effect of High vs Low Dose Intravenous Dexamethasone on Complications in the Immediate Postoperative Phase After Mastectomy- a Randomized, Double-blind, Controlled Trial
Brief Title: High vs Low Dose Dexamethasone on Complications in the Immediate Postoperative Phase After Mastectomy
Acronym: DEX-MAS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Kristin Julia Steinthorsdottir, Principal investigator, MD, Clinical assistant, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DEXMAS01; 2017-000227-27 (EudraCT Number)
Record Dates: First submitted 2017-03-28; First posted 2017-04-24 (Actual); Results first posted 2019-12-02 (Actual); Last update posted 2019-12-02 (Actual); Status verified 2019-11

CONDITIONS: Dexamethasone; Glucocorticoids; Mastectomy; Breast Cancer; Pain, Postoperative; Nausea and Vomiting, Postoperative; Steroid; Systemic Inflammatory Response Syndrome; Postoperative Complications
MeSH Terms: conditions — Breast Neoplasms; Pain, Postoperative; Postoperative Nausea and Vomiting; Systemic Inflammatory Response Syndrome; Postoperative Complications | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexamethasone 8 mg (Active Comparator): Dexamethasone 8 mg pre-operative
  Interventions: Drug: Dexamethasone
- Dexamethasone 24 mg (Active Comparator): Dexamethasone 24 mg pre-operative
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — pre-operative intravenous administration

SUMMARY:
The aim of this study is to investigate the effect of a single preoperative high-dose steroid injection on complications in the immediate postoperative phase after breast cancer surgery, with removal of the breast (mastectomy). Primary outcome is the proportion patients who require transfer to the post anaesthesia care unit (PACU) and the proportion that can be transferred directly to the ward. Secondary outcomes are organospecific complications in the postanesthesia phase, pain and nausea the first 5 days, seroma and wound infection the first 14 days and readmissions the first 30 days after surgery.

The investigators hypothesize that the frequency of transfer to the PACU and organospecific complications will be lower among patients receiving high dose dexamethasone. The investigators hypothesize, that there will be no difference in wound infections, seroma or readmissions.

DETAILED DESCRIPTION:
Post-surgery, patients are traditionally observed and treated in post-anesthesia care units (PACU) until they are discharged to the ward (or directly home) assessed by standardized international discharge criteria.

The research project "Why in PACU?" (Rigshospitalet, Denmark), has since the beginning of 2016 systematically collected and analyzed procedure-related complications in the recovery phase. The complications include pain, nausea/vomiting, circulatory and respiratory problems, orthostatic intolerance and cognitive disorders. Common to all the above-mentioned post-operative problems are the possible links to the inflammatory response caused by the surgical trauma.

Glucocorticoids can in this context be central for the reduction of acute postoperative organ dysfunctions, caused by the anti-inflammatory effect. In a number of different surgical procedures, single dose, pre-operative glucocorticoids have been shown to reduce post-operative nausea and vomiting (PONV), acute pain and need of opioids as well as accelerate the convalescence.

Meta-analyses also showed that single-dose administration of glucocorticoids (methylprednisolone and dexamethasone) for surgical patients is safe as opposed to long-term treatment.

Based on positive results in other procedure-specific studies, all mastectomy patients at Rigshospitalet, have received pre-operative high-dose steroids, in the form of 24 mg dexamethasone injection since mid-2015. This has resulted in a decrease in the proportion of patients who need observation in PACU from 30 % to 10 %. The reduction is primarily due to less pain, less sedation, and lower opioid administration.

Whether this is also partly due to a "systemic effect" (Hawthorn effect) as a result of increased focus on the area cannot be excluded.

Prior to creating clinical recommendations and standards, it is required that the results be tested in a randomized, controlled, clinical trial.

The study is not placebo-controlled since the positive effects of dexamethasone 8 mg on PONV have been shown in numerous trials, and is already being administered to all patients at the clinic. It would therefore not be ethically correct to withdraw from this practise.

ELIGIBILITY:
Inclusion Criteria:

* planned unilateral mastectomy with or without axillary dissection or sentinel node in the study period
* informed signed consent

Exclusion Criteria:

* Chronic/ongoing use of glucocorticoids (except inhalation therapy)
* ongoing use of immunosuppressive therapy
* insulin dependent diabetes
* pregnancy/breastfeeding
* allergies toward study medication, or medication in a standard treatment
* contralateral surgery (lumpectomy/mastectomy) at time of mastectomy
* surgery cannot be performed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2017-03-27 (Actual); Primary Completion 2018-04-22 (Actual); Study Completion 2018-04-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristin J Steinthorsdottir, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No
Not planned to share IPD

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dexamethasone 8 mg | Dexamethasone 24 mg
Started | 65 | 65
Post-randomization Exclusion | 1 (procedure changed, did not receive intervention) | 2 (procedure changed, did not receive intervention)
Completed | 64 | 63
Not Completed | 1 | 2
Not completed — did not receive intervention | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexamethasone 8 mg | Dexamethasone 24 mg | Total
Number analyzed (Participants) | 65 | 65 | 130
Age, Continuous [Mean (Full Range); unit: years] | 66 [28 to 87] | 63 [24 to 85] | 65 [24 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 65 | 128
  Male | 2 | 0 | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Transfer to Post-anesthesia Care Unit (PACU)
Description: Number of patients meeting criteria for transfer to PACU post-surgery
Time Frame: Within 1 hour post-surgery
Population: primary outcome was per intention to treat, secondary outcomes were per protocol (we had 3 post-randomization exclusions, that did not receive the intervention)
Measure: Count of Participants; unit: Participants
Arm/Group | Dexamethasone 8 mg | Dexamethasone 24 mg
Number analyzed (Participants) | 65 | 65
Participants | 23 | 23
Statistical Analysis 1: Comparison: Dexamethasone 8 mg vs Dexamethasone 24 mg; Test type: Superiority; p = 1, Chi-squared; Odds Ratio (OR) = 1.0, 95% CI 2-sided [0.49 to 2.05]

2. Secondary Outcome: Discharge Score,(Modified Aldrete Discharge Score), Operating Room
Description: Danish Society of Anesthesiology and Intensive Care Medicine (DASAIM) discharge score.Construct: The score consists of six modalities (subscores): Sedation,Oxygen saturation,blood pressure,heart rate,pain (at rest)and nausea.Each modality has a score between 0 and 3,and patients are considered dischargeable to the ward when the score sum of all criteria (total score) is 4 or less and no single score is above 1. All values (subscores) are considered best at 0 and worst at 3.
  Sedation: 0 fully awake, 1, sleeping aroused by verbal stimuli, 2 sleeping aroused by physical stimuli, 3 sleeping cannot be aroused.
  Oxygen saturation (%):0 ≥94, 1 90-93, 2 85-89, 3 <85. Blood pressure, systolic (mmHg): 0 100-220, 1 90-99. 2 80-89 or >220, 3<80. Heart rate; pr. min: 0 50-100, 1 101-120, 2 40-49 or 121-130, 3 <40 or >130. Pain (at rest) (Numeric rating scale 0-10): 0 0, 1 0-2, 2 3-6, 3 ≥ 7 Nausea (patient evaluation and nurse observation): 0 none, 1 light, 2 moderate, 3 severe or vomiting.
Time Frame: At transfer from operating room, within 1 hour post-surgery
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Dexamethasone 8 mg | Dexamethasone 24 mg
Number analyzed (Participants) | 63 | 64
score on a scale | 0 [0 to 2] | 1 [0 to 2]
Statistical Analysis 1: Comparison: Dexamethasone 8 mg vs Dexamethasone 24 mg; Test type: Superiority; p = 0.114, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Discharge Score, Arrival at PACU
Description: DASAIM score (Danish Society of Anesthesiology and Intensive Care Medicine). The score consists of six modalities: Sedation, Oxygen saturation, blood pressure, heart rate, pain (at rest) and nausea.
  Each modality has a score between 0 and 3, and patients are considered dischargeable to the ward when the score sum of all criteria is four or less and no single score is above one.
  Sedation: 0 fully awake, 1, sleeping aroused by verbal stimuli, 2 sleeping, aroused by physical stimuli, 3 sleeping, cannot be aroused.
  Oxygen saturation (%): 0 ≥ 94, 1 90-93, 2 85-89, 3 <85. Blood pressure, systolic (mmHg): 0 100-220, 1 90-99. 2 80-89 or >220, 3<80. Heart rate; pr. min: 0 50-100, 1 101-120, 2 40-49 or 121-130, 3 <40 or >130. Pain (at rest) (Numeric rating scale 0-10): 0 0, 1 0-2, 2 3-6, 3 ≥ 7 Nausea (patient evaluation and nurse observation): 0 none, 1 light, 2 moderate, 3 severe or vomiting.
Time Frame: within 3 hours
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Dexamethasone 8 mg | Dexamethasone 24 mg
Number analyzed (Participants) | 63 | 64
score on a scale | 1 [0 to 2] | 1 [0 to 2]
Statistical Analysis 1: Comparison: Dexamethasone 8 mg vs Dexamethasone 24 mg; Test type: Superiority; p = 0.294, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Discharge Score, Arrival at Ward
Description: as for outcome 3
Time Frame: within 3 hours
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Dexamethasone 8 mg | Dexamethasone 24 mg
Number analyzed (Participants) | 63 | 64
score on a scale | 1 [1 to 2] | 1 [1 to 2]

5. Secondary Outcome: Number of Participants With Complication
Description: complications requiring treatment until discharge
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Dexamethasone 8 mg | Dexamethasone 24 mg
Number analyzed (Participants) | 63 | 64
Participants | 12 | 9

6. Secondary Outcome: Total Length of Stay in PACU
Description: Length of stay in the post-anesthesia care unit (PACU), measured as hours and minutes, from start of procedure, to discharge from PACU
Time Frame: 12 hours
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Dexamethasone 8 mg | Dexamethasone 24 mg
Number analyzed (Participants) | 12 | 12
hours | 1.5 [1.4 to 2.4] | 1.5 [1.4 to 1.6]
Statistical Analysis 1: Comparison: Dexamethasone 8 mg vs Dexamethasone 24 mg; Test type: Superiority; p = 0.350, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Total Length of Stay in Hospital
Description: Length of stay in hospital, measured from start of procedure to discharge from hospital to home
Time Frame: 24-48 hours
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Dexamethasone 8 mg | Dexamethasone 24 mg
Number analyzed (Participants) | 63 | 64
hours | 9.2 [7.4 to 24.4] | 11 [8.1 to 23.5]
Statistical Analysis 1: Comparison: Dexamethasone 8 mg vs Dexamethasone 24 mg; Test type: Superiority; p = 0.217, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Secondary Transfer
Description: Secondary transfer to PACU from ward, or to intensive care unit from PACU
Time Frame: 24-48 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Dexamethasone 8 mg | Dexamethasone 24 mg
Number analyzed (Participants) | 63 | 64
Participants | 0 | 0

9. Secondary Outcome: Pain, Numeric Rating Scale
Description: Self-reported pain (worst and average (average through that day), days 0-4) on a numeric rating scale (NRS) 0-10. 0 is no pain, 10 is worst pain imaginable.. Questionnaire.
Time Frame: days 0-4
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Dexamethasone 8 mg | Dexamethasone 24 mg
Number analyzed (Participants) | 52 | 56
score on a scale
  Day 0, average | 2 [0 to 4] | 2 [1 to 4]
  Day 1, average | 2 [0 to 3] | 1 [1 to 2]
  Day 2, average | 1 [0 to 3] | 1 [0 to 2]
  Day 3, average | 1 [0 to 2] | 1 [0 to 1]
  Day 4, average | 1 [0 to 2] | 1 [0 to 1]
  Day 0, worst | 3 [0 to 5.75] | 3 [1 to 5]
  Day 1, worst | 2 [0 to 4] | 1.5 [1 to 3]
  Day 2, worst | 2 [0 to 4] | 2 [0 to 3]
  Day 3, worst | 1 [0 to 1] | 1 [0 to 2]
  Day 4, worst | 1 [0 to 3] | 1 [0 to 2]
Statistical Analysis 1: Comparison: Dexamethasone 8 mg vs Dexamethasone 24 mg; Test type: Superiority; p > 0.193, Wilcoxon (Mann-Whitney) — a priori threshold, bonferroni corrected 0.0125

10. Secondary Outcome: Post Operative Nausea and Vomiting (PONV).
Description: Self-reported nausea, questionnaire, day 0-4. Number of participants reporting nausea and/or vomiting
Time Frame: days 0-4
Measure: Count of Participants; unit: Participants
Arm/Group | Dexamethasone 8 mg | Dexamethasone 24 mg
Number analyzed (Participants) | 52 | 56
Participants
  DAY 0 | 6 | 11
  DAY 1 | 6 | 10
  DAY 2 | 6 | 9
  DAY 3 | 7 | 6
  DAY 4 | 7 | 6
Statistical Analysis 1: Comparison: Dexamethasone 8 mg vs Dexamethasone 24 mg; Test type: Superiority; p > 0.2, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Quality of Sleep
Description: Self-reported quality of sleep (days 0-4). Questionnaire. Dichotomized to Good sleep or sleep problems, numbers reported are number of patients with sleep problems
Time Frame: days 0-4
Measure: Count of Participants; unit: Participants
Arm/Group | Dexamethasone 8 mg | Dexamethasone 24 mg
Number analyzed (Participants) | 52 | 56
Participants
  DAY 0 | 31 | 39
  DAY 1 | 20 | 22
  DAY 2 | 24 | 18
  DAY 3 | 18 | 17
  DAY 4 | 17 | 16
Statistical Analysis 1: Comparison: Dexamethasone 8 mg vs Dexamethasone 24 mg; Test type: Superiority; p > 0.136, Chi-squared

12. Secondary Outcome: Mental Status
Description: Self-reported feelings of restlessness, sadness and fatigue (days 0-4). Questionnaire (anwers possible: yes or no. Numbers are patients answering yes)
Time Frame: days 0-4
Measure: Count of Participants; unit: Participants
Arm/Group | Dexamethasone 8 mg | Dexamethasone 24 mg
Number analyzed (Participants) | 52 | 56
Participants
  DAY 0 : restlessness | 17 | 20
  DAY 0 : sadness | 14 | 18
  DAY 0 : fatigue | 26 | 28
  DAY 1 : restlessness | 9 | 9
  DAY 1 : sadness | 13 | 13
  DAY 1 : fatigue | 11 | 27
  DAY 2 : restlessness | 14 | 8
  DAY 2 : sadness | 14 | 18
  DAY 2 : fatigue | 16 | 17
  DAY 3 : restlessness | 11 | 8
  DAY 3 : sadness | 14 | 20
  DAY 3 : fatigue | 14 | 17
  DAY 4 : restlessness | 13 | 13
  DAY 4 : sadness | 14 | 12
  DAY 4 : fatigue | 14 | 15
Statistical Analysis 1: Comparison: Dexamethasone 8 mg vs Dexamethasone 24 mg; Test type: Superiority; p > 0.003, Chi-squared — A priori threshold for statistical significans was 0.00125 due to multiple comparisons

13. Secondary Outcome: Number of Participants With Seroma, Requiring Treatment
Description: Seroma, requiring treatment the first 14 days.
Time Frame: 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | Dexamethasone 8 mg | Dexamethasone 24 mg
Number analyzed (Participants) | 63 | 64
Participants | 51 | 60
Statistical Analysis 1: Comparison: Dexamethasone 8 mg vs Dexamethasone 24 mg; Test type: Superiority; p = 0.030, Chi-squared; Odds Ratio (OR) = 3.53, 95% CI 2-sided [1.07 to 11.6]

14. Secondary Outcome: Readmission
Description: Any readmission, days 0-30
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Dexamethasone 8 mg | Dexamethasone 24 mg
Number analyzed (Participants) | 63 | 64
Participants | 4 | 4

ADVERSE EVENTS:
Time Frame: 60 hours from administration of study drug
Description: Adverse events are collected from patients that received the study drug (63 and 64 in the 8 and 24 mg group respectively), we had 3 post-randomization exclusion, they did not receive the study drug and adverse events were not collected in agreement with the Good Clinical Practise (GCP) monitor
Arm/Group | Dexamethasone 8 mg | Dexamethasone 24 mg
All-Cause Mortality (participants affected / at risk) | 0/63 | 0/64
Serious Adverse Events (participants affected / at risk) | 5/63 | 3/64
Other Adverse Events (participants affected / at risk) | 0/63 | 0/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dexamethasone 8 mg (N=63) | Dexamethasone 24 mg (N=64)
wound hemorrhage (Surgical and medical procedures) | 5 (5) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-16): https://cdn.clinicaltrials.gov/large-docs/41/NCT03125941/Prot_SAP_000.pdf